CLINICAL TRIAL: NCT06797700
Title: Prediction of Risk Factors of Paraspinal Muscles in Degenerative Lumbar Spondylolisthesis Based on Spine MRI
Brief Title: Risk Factors of Paraspinal Muscles in Degenerative Lumbar Spondylolisthesis
Acronym: RFPMDLS
Status: Not yet recruiting | Type: Observational
Sponsor: The First People's Hospital of Yunnan (Other)
Responsible Party: Principal Investigator, Xinyun li, miss, The First People's Hospital of Yunnan
Other Study IDs: KHLL2025-KY047; 2024JSKFKT-17 (Other Grant/Funding Number: Yunnan Spinal Cord Disease Clinical Medical Center)
Record Dates: First submitted 2025-01-23; First posted 2025-01-28 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-01

CONDITIONS: Spine Degeneration
Keywords: degenerative lumbar spondylolisthesis; paraspinal muscles; MRI

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group A: patients without lumbar spondylolisthesis
- Group B: patients with lumbar spondylolisthesis

SUMMARY:
This is a retrospectively observational study. The goal of this observational study is to analyze the risk factors of paraspinal muscles associated with the occurrence of spondylolisthesis in patients with degenerative lumbar spondylolisthesis(DLS) and to construct a predictive model. The main question it aims to answer is: Which paraspinal muscle changes are risk factors for DLS? We will collect the information of patients who have undergone lumbar MRI in our hospital and have been diagnosed with back pain ( including spondylolisthesis or no spondylolisthesis) during the period from 2022 to 2024.The collected data included gender, age, body mass index (BMI), diabetes, hypertension, occupation and imaging parameters. We will then retrospectively analyze the risk factors associated with lumbar spondylolisthesis.

ELIGIBILITY:
Inclusion Criteria:

* Patients who presented to our hospital with back pain(the diagnosis was spondylolisthesis or no spondylolisthesis);
* Patients older than 50 years;
* Patients with complete clinical data and magnetic resonance imaging (MRI) before surgery.

Exclusion Criteria:

* The patient has previous spinal surgery;
* Patients with lumbar tumor,lumbar infection and lumbar tuberculosis;
* Patients with incomplete MRI sequence.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have undergone lumbar MRI in our hospital and have been diagnosed with back pain ( including spondylolisthesis or no spondylolisthesis) during the period from 2022 to 2024.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-03-06 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
the MF FCSA | Two weeks before treatment
  The functional cross-sectional areas of the multifidus muscl.Measurement it on axial T2-weighted magnetic resonance (MR) images from the L4 vertebral body levels
the ES FCSA | Two weeks before treatment
  The functional cross-sectional areas of the erector spinae.Measurement it on axial T2-weighted magnetic resonance (MR) images from the L4 vertebral body levels
the MF CSA | Two weeks before treatment
  the total cross-sectional areas of the multifidus muscl.Measurement it on axial T2-weighted magnetic resonance (MR) images from the L4 vertebral body levels
the ES CSA | Two weeks before treatment
  the total cross-sectional areas of the erector spinae.Measurement it on axial T2-weighted magnetic resonance (MR) images from the L4 vertebral body levels

SECONDARY OUTCOMES:
SMI | Two weeks before treatment
  The skeletal muscle index.SMI = l CSA of muscle on an axial scan (expressed as cm2) divided by the square of the patient's height (expressed as cm2).

CONTACTS AND LOCATIONS:
Locations (1):
- The First People's Hospital of Yunnan, Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: No